CLINICAL TRIAL: NCT00332670
Title: High Cortisol Levels as a Risk Factor for Depression in the Elderly and the Effect of Bright Light Treatment on Mood, Sleep-Wake Pattern and Self-Sufficiency
Brief Title: Light Therapy for Elderly Depression
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: End of research time, time-resources
Sponsor: GGZ Buitenamstel (Other)
Collaborators: Netherlands Institute for Brain Research, Amsterdam, The Netherlands. (Unknown)
Responsible Party: R. Lieverse, GGZBuitenamstel
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SOW 014-91-049; ZonMw SOW nr 014-91-049; ZonMw AGIKO nr 940-37-033
Record Dates: First submitted 2006-05-31; First posted 2006-06-02 (Estimated); Last update posted 2008-08-15 (Estimated); Status verified 2008-08

CONDITIONS: Major Depressive Disorder
Keywords: (Non-seasonal) Depression; bright light therapy; randomized controlled trial; suprachiasmatic nucleus; HPA-axis; DHEA; melatonin; actigraphy; elderly; self-efficacy; social support
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 10.000lux bright blue light 1hour every morning 1 hour after wake-up time during three weeks
  Interventions: Procedure: 10.000lux blue 1 hour every day during three weeks
- 2 (Placebo Comparator): 50lux dim red light 1 hour every morning 1 hr after wake-up time during 3 weeks
  Interventions: Procedure: 50lux dim red 1 hour every day during three weeks

INTERVENTIONS:
Procedure: 10.000lux blue 1 hour every day during three weeks — 10.000lux during 60 minutes, starting 1 hour after wake-up, during 3 weeks
  Other Names: Bright light
  Arms: 1
Procedure: 50lux dim red 1 hour every day during three weeks — 50 lux red light, 60 minutes every morning, starting 1 hour after wake-up, during three weeks
  Other Names: Dim red light
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the following two hypotheses:

1. Treatment with bright light improves their sleep, mood, concentration and self-sufficiency of elderly depressed subjects. This clinical improvement is accompanied by decreases in cortisol/DHEA ratio and increases in melatonin concentration in urine and saliva.
2. The eventual beneficial effect of bright light treatment can be predicted by the presence of sleep-wake rhythm disturbances as found using muscle activity registration, and by cortisol/DHEA and melatonin concentrations in saliva and urine over the day and the night.

DETAILED DESCRIPTION:
Background: Depression frequently occurs in the elderly. In normal aging, and in depression, the functioning of the suprachiasmatic nucleus (SCN) is impaired, as evidenced by an increased prevalence of day-night rhythm perturbations, e.g. sleeping disorders. Also, the normal inhibition of SCN neurons on corticotrophin-releasing hormone (CRH) producing cells is decreased, which could be responsible for the hyperactive hypothalamus-pituitary adrenocortical axis (HPA-axis). This raises the question whether elderly patients with depression have more impaired SCN activity and whether HPA-activity is enhanced. Using bright light therapy (BLT) the SCN can be stimulated. And, the beneficial effects of BLT on seasonal depressive disorders are well accepted. Nevertheless, the effects of BLT in aged depressed patients have never been studied, as yet.

Aims: The aim of this study is to test the hypothesis that BLT improves sleep, mood, concentration and self-efficacy of older people with depression and this improvement is accompanied by a normalization of HPA-indices.

Methods: Randomised double blind placebo controlled trial in 120 subjects of 60 years and older with a diagnosis of major depressive disorder (DSM-IV/SCID-I). Subjects are recruited through referrals of psychiatric outpatient clinics and from case-finding from databases of general practitioners and old-people homes in the Amsterdam region. After inclusion subjects are randomly allocated to bright blue light vs. dim red light groups using two Philips Bright Light Energy boxes type HF 3304 per subject from which the light bulbs have been covered with bright blue or dim red light permitting filters. Criteria for stratification are the use of SSRIs. Prior to treatment a 1-week run-in period without treatment will be used as a baseline condition. At three time points several endocrinological, psychophysiological, psychometrically, neuropsychological, and neuroimaging measures are performed: just before start of light therapy (T0), after completion of the three week light therapy period (T1), and three weeks thereafter (T2).

Relevance: This study is designed to show whether light therapy can reduce depressive symptoms of elderly patients with a major depressive disorder. If this is the case, then additional lightning may easily be installed in the homes of patients to serve as a maintenance treatment. Also, if our data support the role of a dysfunctional biological clock in depressed elderly subjects, such a finding may guide the further development of drugs that inhibit the HPA axis.

ELIGIBILITY:
Inclusion Criteria:

* Understanding and speaking Dutch language
* 60 years of age or older
* Presence of a Major Depressive Disorder according to DSM-IV (SCID-based)
* When under treatment of an ophthalmologist, his / her approval for participation.

Exclusion Criteria:

* Progressive eye diseases, glaucoma or cataract for which an operation is scheduled in near future, aphakia, retinopathies like maculopathy, retinitis pigmentosa or ablatio retina.
* Physical problems or disorders which require specific medical treatment like Lupus, untreated diabetes, malignancies, organic brain disorders, chronic infections, thyroid disorders not adequately treated, thyroid associated ophthalmopathies, M. Parkinson.
* Presence of any concurrent substance abuse problem
* Presence of other actual axis-I disorders like bipolar disorder, dementias, delirium, all psychotic disorders, Posttraumatic stress disorder.
* Use of tricyclic antidepressants, MAOIs.
* Use of corticosteroids.
* Use of tetracyclic antibiotics.
* Treatment with antidepressants shorter than 2 months
* Use of oral contraceptives.
* Treatment with light therapy in the past.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2003-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HADRS-17) | at T0, T1 and T2

SECONDARY OUTCOMES:
Actimetry | continuous measurement during complete 7 week study period
24-hour urinary cortisol measurements | at T0, T1 and T2 (saliva melatonin evening curve (bedtime minus 4 hours, minus 3 hours, minus 2 hours, minus 1 hour).
saliva cortisol daytime curve | T0, T1 and t2 (get-up time plus 30 minutes, plus 60 minutes, plus 90 minutes, plus 120 minutes,bedtime minus 4 hours, minus 3 hours, minus 2 hours, minus 1 hour)
Social Rhythm Metric | complete 7-week study period.
Groningen Activity Restriction Scale (GARS) | at T0, T1 and T2
Algemene Competentieverwachtingen Schaal (ALCOS) | at T0, T1 and T2
Social Support List interactions, discrepancies and negative (SSL-i, SSL-d, SSL-n) | at T0, T1 and T2
MOS-short form General Health Survey (SF-20) | T0, T1 and T2
Pittsburgh Sleep Quality Inventory (PSQI) | at T0, T1 and T2
Neuropsychological test battery | at T0, T1 and T2
fMRI (encoding task, recognition task, N-Back) | at T0 and T1
structural MRI scanning (brain and volumetry of adrenals) | at T0 and T1
MADRS | at T0, T1 and t2
Adverse effects inventarisation | 3-5 times during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Witte JG Hoogendijk, prof. dr., Study Director — Center for Neurogenomics and Cognitive Research, Free University, Amsterdam, the Netherlands; Department of Psychiatry VU University Medical Center, Amsterdam, The Netherlands; GGZ Buitenamstel, Amsterdam, The Netherlands; Eus van Someren, PhD, Study Chair — Netherlands Institute for Brain Research, Amsterdam, The Netherlands; VU University Medical Center, Amsterdam, The Netherlands; Marjan MA Nielen, PhD, Study Chair — Center for Neurogenomics and Cognitive Research, Free University, Amsterdam, the Netherlands; Department of Psychiatry VU University Medical Center, Amsterdam, The Netherlands; GGZ Buitenamstel, Amsterdam, The Netherlands; Ritsaert Lieverse, MD, Principal Investigator — Center for Neurogenomics and Cognitive Research, Free University, Amsterdam, the Netherlands; Department of Psychiatry VU University Medical Center, Amsterdam, The Netherlands; GGZ Buitenamstel, Amsterdam, The Netherlands
Locations (1):
- GGZ Buitenamstel, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Background] Hoogendijk WJ, van Someren EJ, Mirmiran M, Hofman MA, Lucassen PJ, Zhou JN, Swaab DF. Circadian rhythm-related behavioral disturbances and structural hypothalamic changes in Alzheimer's disease. Int Psychogeriatr. 1996;8 Suppl 3:245-52; discussion 269-72. doi: 10.1017/s1041610297003426. No abstract available. PMID 9154571
- [Background] Beekman AT, Penninx BW, Deeg DJ, Ormel J, Braam AW, van Tilburg W. Depression and physical health in later life: results from the Longitudinal Aging Study Amsterdam (LASA). J Affect Disord. 1997 Dec;46(3):219-31. doi: 10.1016/s0165-0327(97)00145-6. PMID 9547118
- [Background] Deuschle M, Gotthardt U, Schweiger U, Weber B, Korner A, Schmider J, Standhardt H, Lammers CH, Heuser I. With aging in humans the activity of the hypothalamus-pituitary-adrenal system increases and its diurnal amplitude flattens. Life Sci. 1997;61(22):2239-46. doi: 10.1016/s0024-3205(97)00926-0. PMID 9393943
- [Background] Kripke DF, Tuunainen A, Endo T. Benefits of light treatment for depression. Am J Psychiatry. 2006 Jan;163(1):162-3; author reply 163. doi: 10.1176/appi.ajp.163.1.162-b. No abstract available. PMID 16390913
- [Background] Kripke DF. Light treatment for nonseasonal depression: speed, efficacy, and combined treatment. J Affect Disord. 1998 May;49(2):109-17. doi: 10.1016/s0165-0327(98)00005-6. PMID 9609674
- [Background] Golden RN, Gaynes BN, Ekstrom RD, Hamer RM, Jacobsen FM, Suppes T, Wisner KL, Nemeroff CB. The efficacy of light therapy in the treatment of mood disorders: a review and meta-analysis of the evidence. Am J Psychiatry. 2005 Apr;162(4):656-62. doi: 10.1176/appi.ajp.162.4.656. PMID 15800134
- [Background] Wirz-Justice A, Terman M, Oren DA, Goodwin FK, Kripke DF, Whybrow PC, Wisner KL, Wu JC, Lam RW, Berger M, Danilenko KV, Kasper S, Smeraldi E, Takahashi K, Thompson C, van den Hoofdakker RH. Brightening depression. Science. 2004 Jan 23;303(5657):467-9. doi: 10.1126/science.303.5657.467c. No abstract available. PMID 14739440
- [Background] Wirz-Justice A, Benedetti F, Berger M, Lam RW, Martiny K, Terman M, Wu JC. Chronotherapeutics (light and wake therapy) in affective disorders. Psychol Med. 2005 Jul;35(7):939-44. doi: 10.1017/s003329170500437x. PMID 16045060
- [Background] Martiny K, Lunde M, Unden M, Dam H, Bech P. Adjunctive bright light in non-seasonal major depression: results from clinician-rated depression scales. Acta Psychiatr Scand. 2005 Aug;112(2):117-25. doi: 10.1111/j.1600-0447.2005.00574.x. PMID 15992393
- [Background] Martiny K, Lunde M, Unden M, Dam H, Bech P. Adjunctive bright light in non-seasonal major depression: results from patient-reported symptom and well-being scales. Acta Psychiatr Scand. 2005 Jun;111(6):453-9. doi: 10.1111/j.1600-0447.2005.00532.x. PMID 15877712
- [Background] Gordijn MC, Beersma DG, Korte HJ, Van den Hoofdakker RH. Testing the hypothesis of a circadian phase disturbance underlying depressive mood in nonseasonal depression. J Biol Rhythms. 1998 Apr;13(2):132-47. doi: 10.1177/074873098128999989. PMID 9554575
- [Background] Zhou JN, Riemersma RF, Unmehopa UA, Hoogendijk WJ, van Heerikhuize JJ, Hofman MA, Swaab DF. Alterations in arginine vasopressin neurons in the suprachiasmatic nucleus in depression. Arch Gen Psychiatry. 2001 Jul;58(7):655-62. doi: 10.1001/archpsyc.58.7.655. PMID 11448372
- [Derived] Lieverse R, Van Someren EJ, Nielen MM, Uitdehaag BM, Smit JH, Hoogendijk WJ. Bright light treatment in elderly patients with nonseasonal major depressive disorder: a randomized placebo-controlled trial. Arch Gen Psychiatry. 2011 Jan;68(1):61-70. doi: 10.1001/archgenpsychiatry.2010.183. PMID 21199966
- [Derived] Lieverse R, Nielen MM, Veltman DJ, Uitdehaag BM, van Someren EJ, Smit JH, Hoogendijk WJ. Bright light in elderly subjects with nonseasonal major depressive disorder: a double blind randomised clinical trial using early morning bright blue light comparing dim red light treatment. Trials. 2008 Jul 31;9:48. doi: 10.1186/1745-6215-9-48. PMID 18671864